CLINICAL TRIAL: NCT04973384
Title: Ocular Comorbidity in Atopic Dermatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Pernille Rævdal, MD, PhD-student, Coordinating researcher,, Rigshospitalet, Denmark
Other Study IDs: H-20069664
Record Dates: First submitted 2021-07-06; First posted 2021-07-22 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Atopic Keratoconjunctivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collection of tear samples, brush swabs and conjunctival imprints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A clinical characterization of a large cohort of patients with different severities of AD and ocular symptoms/atopic keratoconjunktivitis (AKC). The data will contribute to assess the frequency of complications in order to give a rationale for focused prevention and treatment strategy.

DETAILED DESCRIPTION:
Atopic Dermatitis (AD), a very common inflammatory skin condition of child and adulthood, is strongly associated with ocular disease. Accordingly, about 20% experience conjunctivitis at some point, and many have chronic disease. Atopic keratoconjunctivitis (AKC) is the most feared as it may lead to blindness. Little is known about the etiology, the immune infiltrate, as well as predictive factors of AKC and the clinical characteristics of AD patients who develop this entity. We expect this project to enable clinicians to better identify AKC patients in the future as well as improve the understanding of the pathogenesis of AKC.

The ocular findings will be compared between AD severity and a control group without ocular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Danish talking
* Diagnosed with atopic dermatitis (AD)
* Current or previous ocular symptoms suspected to be atopic keratoconjunctivitis

Exclusion Criteria:

* No pause in eyedrops
* Ocular infections within the last 3 months
* Use of local or systemic antibiotics within the last 3 months
* Significant untreated systemic disease such as hypertension, heart failure, diabetes mellitus, previous cerebral infarction or bleeding, lung diseases and autoimmune diseases other than atopic dermatitis and related comorbidities. The diseases are accepted if they are well treated or do not require treatment
* Current pregnant or breastfeeding
* Use of contact lenses, unless these are paused 2 weeks before the examination or they are due to keratoconus treatment
* If the eye symptoms turn out not to be related to atopic keratoconjunctivitis
* If it is assessed that the individual cannot participate sufficiently for the examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AD patients with current or previous ocular symptoms suspected to be atopic keratoconjunctivitis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bulbar redness (BR) score | 1 day At examination
  Difference in Bulbar redness (BR) score (Keratograph 5M, R-scan). Scale from 0-4. A higher score indicates more severe BR.

SECONDARY OUTCOMES:
Inferior Tear Meniscus Height (TMH) | 1 day Cross-sectional at examination (one time)
  Difference in Inferior Tear Meniscus Height (TMH) (Keratograph 5M)
Non-invasive Keratograph Break-Up Time (NIKBUT) | 1 day Cross-sectional at examination (one time)
  Difference in Non-invasive Keratograph Break-Up Time (NIKBUT) (Keratograph 5M)
Meibo-Scan | 1 day Cross-sectional at examination (one time)
  Difference in Meibo-Scan (Keratograph 5M). Scale from 0-3. A higher score indicates more morphological changes.
Ocular surface staining | 1 day Cross-sectional at examination (one time)
  Difference in Ocular surface staining
Osmolarity of the tears | 1 day Cross-sectional at examination (one time)
  Difference in Osmolarity of the tears (TearLab™)
Fluorescein tear break up time (TFBUT) | 1 day Cross-sectional at examination (one time)
  Difference in Fluorescein tear break up time (TFBUT)
Schirmer's I test | 1 day Cross-sectional at examination (one time)
  Difference in Schirmer's I test
Intraocular pressure (IOP) | 1 day Cross-sectional at examination (one time)
  Difference in Intraocular pressure (IOP)
Pentacam investigations for detection of keratoconus | 1 day Cross-sectional at examination (one time)
  Difference in the frequency of keratoconus
Tear cytokine analysis | 1 day Cross-sectional at examination (one time)
  Difference in the levels of inflammatory cytokines in the tears
Tear proteomic analysis | 1 day Cross-sectional at examination (one time)
  Difference in the protein profile in the tears
Tear MUC5AC analysis | 1 day Cross-sectional at examination (one time)
  Difference in the level of MUC5AC in tears
Goblet cell density | 1 day Cross-sectional at examination (one time)
  Difference in goblet cells density
Microbiome analysis | 1 day Cross-sectional at examination (one time)
  Difference in the amount of different species of the Microbiome of the ocular surface
Investigation of the infestation of Demodex | 1 day Cross-sectional at examination (one time)
  Difference in the amount of Demodex mites in the eyelashes/eyelids with non-invasive in vivo confocal microscopy
OSDI-score | 1 day Cross-sectional at examination (one time)
  Difference in the Ocular Surface Disease Index (OSDI) score. A 12-item questionnaire that gives a score on a scale from 0 to 100, where higher scores represent greater disability (mild [13-22 points], moderate [23-32 points], and severe [33-100 points]).
PO-SCORAD | 1 day Cross-sectional at examination (one time)
  Difference in the Patient-Oriented SCORing of Atopic Dermatitis (POSCORAD) score. A validated self-assessment tool to clinical evaluate AD severity, using subjective and objective criteria. A higher score indicates more severe AD.
POEM | 1 day Cross-sectional at examination (one time)
  Difference in the Patient Oriented Eczema Measure (POEM) score. A validated self-assessment tool to clinical evaluate AD severity. A scale from 0-28. A higher score indicates more severe AD.
EASI | 1 day Cross-sectional at examination (one time)
  Difference in Eczema Area and Severity Index (EASI) score. A tool used to measure the extent (area) and severity of atopic eczema. A scale from 0-72. A higher score indicates more severe AD.
best-corrected logMAR acuity | 1 day Cross-sectional at examination (one time)
  Difference in best-corrected logMAR acuity
Slit lamp examination | 1 day Cross-sectional at examination (one time)
  Difference in observations with slit lamp

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Heegaard, MD, DMSci, Principal Investigator — Department of Ophthalmology, Rigshospitalet-Glostrup
Locations (1):
- Department of Ophthalmology, Rigshospitalet-Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No